CLINICAL TRIAL: NCT04523064
Title: Empagliflozin for Prevention of Acute Kidney Injury in Patients With Type 2 Diabetes Mellitus Undergoing Extracorporeal On-pump CABG: The POST-CABGDM Trial
Brief Title: POST-CABGDM: Empagliflozin in Perioperative CABG
Acronym: POST-CABGDM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4957/19/176
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 2; Coronary Artery Disease; Coronary Artery Bypass Surgery; Acute Kidney Injury
Keywords: Diabetes; Coronary artery disease; SGLT2i; CABG; Acute kidney injury
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease; Acute Kidney Injury; Diabetes Mellitus | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SGLT2i (empagliflozin) (Active Comparator): Empagliflozin 25 mg 1 time day for three months
  Interventions: Drug: Empagliflozin 25 MG
- Standard of care (No Intervention): Standard care treatment of diabetes patients in our center

INTERVENTIONS:
Drug: Empagliflozin 25 MG — Patients with diabetes waiting for surgery will receive empagliflozin for at least three months.
  Other Names: Jardiance 25 mg
  Arms: SGLT2i (empagliflozin)

SUMMARY:
Introduction: Diabetes Mellitus (DM) is a condition known to be associated with coronary artery disease (CAD) and its role as promoter of atherosclerosis is well stablished. The revascularization surgery is commonly indicated to patients with multivessel coronary disease and kidney injury is a prevalent complication in post operation. This work aims to evaluate the impact of a strategy to control Diabetes Mellitus using inhibitors of sodium-glucose cotransporters (ISGLT2) in diabetics patients with assigned myocardial revascularization with cardiopulmonary bypass

DETAILED DESCRIPTION:
Random Prospective Study non-blinded with 144 diabetics patients designated to myocardial revascularization with cardiopulmonary bypass . 72 patients will be randomly set to usual treatment provided by health care service and 72 patients will be randomly assigned treatment based on ISGLT2 (Empaglifozin). Patients will receive treatment as set for 3 months until 3 days prior to surgery. Creatinine levels will be measured immediately after surgery and in the following 3 days in post-op.

To evaluate the possibility to reduce the acute kidney injury in a randomized group treated with therapy based on ISGLT2.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Type 2 diabetes mellitus
* Multivessel CAD documented by coronary angiography with formal indication for CRM.

Exclusion Criteria:

* eGFR <30mL / min / 1.73m2 or dialysis therapy;
* Inability to sign the informed consent form;
* Contraindication to CABG on pump;
* Need for urgent or emergency CABG;
* Terminal or disabling illness with reduced life expectancy;
* Pregnancy in progress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | 3 months
  Development of post-CABG acute kidney injury according to RIFFLE or AKIN or KDIGO criteria

SECONDARY OUTCOMES:
Atrial fibrillation | 3 months
  Development of atrial fibrillation during hospital admission
Pulmonary infection | 3 months
  Development of pulmonary infection during hospital admission
Infection of surgical site | 3 months
  Development of infection of surgical site during hospital admission
ICU readmission | 3 months
  Transfer to ICU during hospital admission
Need for IV insulin | 3 months
  Need for IV insulin during hospital admission
Myocardial Infarction Type 5 | 3 months
  Occurence of myocardial infarction type 5 during admission

CONTACTS AND LOCATIONS:
Overall Officials: Carlos V Serrano, MD, PhD, Principal Investigator — Instituto do Coração - Hospital das Clinicas FMUSP
Locations (1):
- University of Sao Paulo Medical School - The Heart Institute, São Paulo, São Paulo, Brazil